CLINICAL TRIAL: NCT01390350
Title: A Multi-center, Double-blind, Placebo-controlled Phase II Study of the Efficacy and Safety of Canakinumab in Subjects With Schnitzler Syndrome
Brief Title: Ilaris® Effects in Schnitzler Syndrome (ILESCH)
Acronym: ILESCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Karoline Krause, Karoline Krause, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CACZ885DDE03T; 2010-024156-28 (EudraCT Number)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Schnitzler Syndrome
Keywords: Schnitzler syndrome; autoinflammatory syndrome
MeSH Terms: conditions — Schnitzler Syndrome | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Canakinumab (Experimental)
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab — 150mg subcutaneous injections on day 0
  Other Names: Ilaris
  Arms: Canakinumab
Drug: Placebo — 150mg subcutaneous injections on day 0
  Arms: Placebo

SUMMARY:
This is a multi-center double-blind placebo-controlled study to assess the efficacy and safety of canakinumab (trade name Ilaris®), a high-affinity monoclonal antibody that neutralizes IL-1β, in patients with Schnitzler syndrome. Efficacy is assessed by physician's global assessment (a combined clinical symptom score) and inflammation markers. Following a baseline period of 1-4 weeks, patients will be randomized to receive single s.c. injections of either 150 mg canakinumab or placebo (day 0). Treatment response will be assessed on day 7. Patients will then be eligible to enter the 16-week open-label phase and receive canakinumab injections (150-300mg, dose depends on clinical response on day 7) upon relapse of symptoms. Visits for investigator's assessments will be scheduled at 4-weekly intervals following day 7. Overall a max. of 20 subjects with Schnitzler syndrome will be enrolled.

1. Amendment: After successful completion of the 16-week open-label phase patients will be eligible to enter a one-year open-label extension of the study. During this part of the study patients will be scheduled at bi-monthly intervals. Canakinumab dosing will be performed upon relapse of symptoms comparable to the 16-week open-label phase.
2. Amendment: After successful completion of the 1-year open-label study extension patients will be eligible to enter another 3-year open-label extension. Patients will be scheduled at 3-month-intervals and Canakinumab dosing will be performed on an individual basis with optimized dosing intervals to ensure a constant low disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Informed consent signed and dated
* Able to read, understand and willing to sign the informed consent form and abide with study procedures
* SchS diagnosis based on diagnostic criteria defined in Appendix
* Patients with symptomatic Schnitzler syndrome [SchS] (as defined by the physician's global assessment with a minimum score of 8 and C-reactive protein [CRP] > upper limit of normal [ULN])
* Willing, committed and able to return for all clinic visits and complete all study-related procedures, including willingness to have subcutaneous injections administered by a qualified person
* In females of childbearing potential: Negative pregnancy test; females willing to use highly effective contraception (Pearl-Index < 1). A woman will be considered not of childbearing potential if she is post-menopausal for greater than two years or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy)
* Subjects are considered eligible, if they meet the following tuberculosis [TB] screening criteria: no history of latent or active TB prior to screening, no signs or symptoms suggestive of active TB, no recent close contacts with a person with active TB, and negative QuantiFERON-TB test at screening (if QuantiFERON-TB test is positive, the patient can only be included if active TB is ruled out with appropriate measurements according to standard of care)
* No participation in other clinical trials 4 weeks before and after participation in this study

Exclusion Criteria:

* Concurrent/ongoing treatment with anakinra (Kineret®) or recent treatment within 48 hours prior to day 0
* Concurrent/ongoing treatment with other biologics or recent treatment (less than 5 half lives)
* Concurrent/ongoing treatment with immunosuppressives (e.g. cyclosporine, methotrexate, dapsone or others) within 4 weeks or 5 half lives prior to day 0, whichever is longer
* Concurrent/ongoing treatment with high doses of systemic steroids (>20mg prednisolone equivalent)
* Evidence of recurrent or latent systemic infection such as TB
* Significant medical condition rendering the patient immunocompromised or not suitable for a clinical trial
* Treatment with a live (attenuated) virus vaccine during three months prior to day 0 and for 3 months after end of study
* Evidence of tuberculosis as defined by local guidelines/ local medical practice (at screening)
* An abnormal chest radiograph consistent with clinical signs of prior or present tuberculosis infection whether or not previously treated with anti-tuberculosis agents
* A history of listeriosis, active persistent chronic or active infection(s) requiring treatment with parenteral antibiotics, parenteral antivirals, or parenteral antifungals within four weeks prior to day 0
* Significant concomitant illness that would adversely affect the subject's participation or evaluation in this study
* Evidence of current HIV, active hepatitis B, or hepatitis C infection by serological screening
* History of malignancies within five years prior to screening other than a successfully treated non-metastatic cutaneous, basal, or squamous cell carcinoma and/or in situ cancer
* Presence of any of the following laboratory abnormalities at enrollment visit: creatinine >2.0 x ULN, WBC <3000/µl; platelet count <100000/µl ; alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >3.0 x ULN
* Lactating females or pregnant females
* Subjects for whom there is concern about compliance with the protocol procedures
* Any medical condition which, in the opinion of the Investigator, would interfere with participation in the study or place the subject at risk
* History of substance abuse (drug or alcohol) or any other factor (e.g., serious psychiatric condition) within the last 5 years that could limit the subject's ability to comply with study procedures
* Subjects who are detained officially or legally to an official institute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2017-12-21 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The effect of canakinumab on the clinical signs and symptoms of SchS measured by physician's global assessment | 16 months
  Proportion of patients with complete response (based on physician's global assessment on overall autoinflammatory disease activity) at day 7 in the canakinumab treated group as compared to the placebo group

SECONDARY OUTCOMES:
The safety and tolerability of canakinumab in subjects with Schnitzler syndrome | 16 months
The change in biomarkers of inflammation during the treatment period with canakinumab | 16 months
  Biomarkers of inflammation include C-reactive protein, serum amyloid A and erythrocyte sedimentation rate
Changes in patients' quality of life during the treatment period with canakinumab | 16 months
  Patient's quality of life assessment includes the Dermatology Life Quality Index and SF 36

CONTACTS AND LOCATIONS:
Overall Officials: Karoline Krause, MD, Principal Investigator — Charité University, Berlin
Locations (5):
- Germany (5):
  - Allergie-Centrum-Charité, Charité University, Berlin
  - Dept. of Dermatology, Klinikum Darmstadt, Darmstadt
  - Dept. of Dermatology, University Heidelberg, Heidelberg
  - Dept. of Dermatology, University Münster, Münster
  - Dept. of Dermatology, University Tübingen, Tübingen